CLINICAL TRIAL: NCT04726670
Title: Effect of EDDY and Manual Dynamic Activation Techniques on Postoperative Pain in Retreatment: a Randomized Controlled Trial
Brief Title: Effect of EDDY and Manual Dynamic Activation Techniques on Postoperative Pain in Retreatment
Acronym: Pain
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-549
Record Dates: First submitted 2021-01-23; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A Comparison of Pain Levels: A Comparison of Pain Levels at different time intervals according to the Irrigation Activation Protocols
  Interventions: Other: Evaluation of postoperative pain
- The evaluation of postoperative pain (Mean Rank) within the group according to time periods: The evaluation of postoperative pain (Mean Rank) within the group according to time periods
  Interventions: Other: Evaluation of postoperative pain

INTERVENTIONS:
Other: Evaluation of postoperative pain — A participant voluntary consent form was obtained from each patient. Ninety patients were numerically coded in computer environment by someone who was not included in the study for randomization (www.random.org).
  A single clinician performed retreatment on each of the 90 teeth during a single visit.

SUMMARY:
The aim of the study was to evaluate the effectiveness of EDDY and manual dynamic activation (MDA) techniques on postoperative pain (PP) associated in retreatment. Ninety patients scheduled for retreatment were treated at one visit. After the single visit retreatment procedure, the patients were divided into two groups (n = 45) on the basis of the need for additional irrigation activation procedures (EDDY and MDA). The patients' post-treatment pain levels were asked to rate the intensity of their pain on a 10-point numerical rating scale (NRS) at 12th, 24th, 48th, and 72th hours and 7 days.

DETAILED DESCRIPTION:
The sample size was based on pilot study data that indicated that 38 patients would be sufficient for each group (type I alpha error = 5%, effect size = 0.7, power = 80%). To compensate for possible dropouts during the treatment and/or follow-up periods, 45 patients were assigned to each group.The study protocol was approved by the Ankara Yıldırım Beyazıt University Ethical Board of Clinical Trials and Non-interventional Research (2019-549).The inclusion criteria were as follows:

1. Healthy individuals aged 18 to 40 years.
2. Devital mandibular premolar teeth with asymptomatic periapical lesions.
3. Teeth with initial root canals filled 2-4 mm short of the apex.
4. Premolar teeth with periapical radiolucency (PAI 3-4) [12] detected by radiographic examination.
5. Coronal restoration.
6. Teeth on which root canal treatment had been performed in the researcher's hospital at least 4 years prior to the study.

The exclusion criteria were as follows:

1. The use of drugs, such as analgesics, anti-inflammatories, and antibiotics, for pain and infection control in the previous 12 hours.
2. A history of susceptibility or adverse reactions to any drugs or materials used in the study.
3. Teeth with open apexes and resorption.
4. Teeth with post-core restoration.
5. Vertical root fractures and teeth on which surgery had been performed.
6. Pregnancy and breastfeeding. A participant voluntary consent form was obtained from each patient. Ninety patients were numerically coded in computer environment by someone who was not included in the study for randomization (www.random.org)A single clinician performed retreatment on each of the 90 teeth during a single visit. A 27-gauge dental injector (Set Inject; Set Medical Instruments, Istanbul, Turkey) was used to anesthetize the patients with a solution of 40 mg Articain and 0.006 mg/mL epinephrine (Ultracain DS Forte; Aventis, Istanbul, Turkey). Old restorations and caries were removed, and on the basis of the straight-line principle, round diamond burs were used to create access cavities under rubber dam isolation. All subsequent treatment procedures were performed under rubber dam isolation, and 3.5× (Zumax Sle Loupe) magnification was used. When necessary, the cervical margin was elevated with composite resin to ensure the continuity of the isolation.

The gutta-percha and sealer were removed with hand files and ProTaper retreatment (Dentsply Maillefer) files. No solvent was used. The working length was calculated with a ProPex Pixi apex locater (Dentsply Maillefer). Periapical radiography allowed for the calculation of the working length and confirmation of the removal of the previous canal filling. Root canals were enlarged to be ProTaper Universal F3 (30/0.9). A lubricant (Glyde File Prep, Dentsply DeTrey, GmbH, Konstanz, Germany) was used between each file to prevent the rotary files from getting stuck in the root canal. A total of 20 mL 2.5% sodium hypochlorite (NaOCl) irrigation solution (Werax, Izmir, Turkey) was used for each treatment. For all teeth, the final irrigation was performed with 5 mL 17% ethylenediaminetetraacetic acid (EDTA) solution (Werax, Izmir, Turkey) for 1 minute. After the retreatment procedure, the patients were divided into two groups on the basis of the additional irrigation activation procedures with 6 mL 2.5% NaOCl (n = 45). Information on which irrigation activation methods to use was not given to the patient.

First group (manual dynamic activation): A final rinse with 6 mL 2.5% NaOCl was done performed after shaping, using a ProTaper Universal F3 (Dentsply, Maillefer, Ballaigues, Switzerland) gutta-percha up and down movements to as 1 mm short from the working length for 1 minute.

Second group (EDDY): A 28 mm long polyamide tip with 25.04 taper was adapted to TA-200 (Micron, Tokyo, Japan) and operated at 6,000 Hz, the maximum speed setting. It was placed in the canal 2 mm shorter than the working length. Next, 6 mL 2.5% NaOCl was administered to the canal in three 20-second activation-nonactivation cycles (2 ml/20 seconds).

The root canals were dried with paper points (Dentsply, Sirona). The working length was reached with ProTaper Universal F3 gutta-percha (Dentsply, Sirona), and tug-back was taken. The gutta-percha was covered with a sealer (AH Plus; Dentsply, Sirona), and root canal fillings were performed with a single-cone technique. After the completion of the root canal filling procedures, the residual materials were removed with a heat source. A resin composite (3M, ESPE) was used for the coronal restorations. Occlusal reduction was performed on all the teeth included in the study. No antibiotics or analgesics were prescribed.

Patient questionnaire The postoperative follow-up and evaluation of the cases were performed by a researcher who had no knowledge of the study group. A 10-point numerical rating scale (NRS) was introduced to the patients, and they were asked to rate their post-treatment pain by telephone after 12, 24, 48, and 72 hours. The antibiotics and analgesics were questioned. The patients were called for clinical examination 1 week later. Palpation and percussion sensitivity in the treated teeth was determined on the basis of the patients' perceptions of pain. All percussion tests were performed by the same operator to ensure standardization. The measurement values were based on the 10-point NRS. The pain scores were placed into the following four categories: 0 = none, 1-3 = mild, 4-6 = moderate, and 7-10 = severe.

ELIGIBILITY:
Inclusion Criteria:

- 1- Healthy individuals aged 18 to 40 years. 2- Devital mandibular premolar teeth with asymptomatic periapical lesions. 3- Teeth with initial root canals filled 2-4 mm short of the apex. 4- Premolar teeth with periapical radiolucency (PAI 3-4) [12] detected by radiographic examination.

5- Coronal restoration. 6- Teeth on which root canal treatment had been performed in the researcher's hospital at least 4 years prior to the study.

Exclusion Criteria:

* 1- The use of drugs, such as analgesics, anti-inflammatories, and antibiotics, for pain and infection control in the previous 12 hours.

  2- A history of susceptibility or adverse reactions to any drugs or materials used in the study.

  3- Teeth with open apexes and resorption. 4- Teeth with post-core restoration. 5- Vertical root fractures and teeth on which surgery had been performed. 6- Pregnancy and breastfeeding.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients referred to the endodontic clinic for retreatment were asked to complete a questionnaire to provide pre-treatment clinical conditions and demographic data. participant voluntary consent form was obtained from each patient. Ninety patients were numerically coded in computer environment by someone who was not included in the study for randomization (www.random.org).
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
Effect of EDDY and manual dynamic activation techniques on postoperative pain in retreatment: a randomized controlled trial | 1.5 years
  Evaluation of postoperative pain

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yildirim BEYAZIT UNIVERSITY, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gundogar M, Sezgin GP, Kaplan SS, Ozyurek H, Uslu G, Ozyurek T. Postoperative pain after different irrigation activation techniques: a randomized, clinical trial. Odontology. 2021 Apr;109(2):385-392. doi: 10.1007/s10266-020-00553-5. Epub 2020 Sep 11. PMID 32915346
- [Derived] Ince-Yusufoglu S, Keskin NB, Uslu G, Helvacioglu-Yigit D. Effect of EDDY and manual dynamic activation techniques on postoperative pain in non-surgical retreatment: a randomized controlled trial. BMC Oral Health. 2023 Jan 3;23(1):3. doi: 10.1186/s12903-022-02702-4. PMID 36597145